CLINICAL TRIAL: NCT00142740
Title: Population Genetics and Immune Response to Hepatitis B Vaccination in Adolescents: A Substudy of ATN 024 and ATN 025
Brief Title: Hepatitis B Vaccine Genetics: A Substudy of ATN 024 and ATN 025
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 052
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: HIV Infection; Hepatitis B
Keywords: Hepatitis B vaccines; HIV-infected adolescents; Hepatitis B infection (negative); HIV vaccine trial
MeSH Terms: conditions — HIV Infections; Hepatitis B

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 5 ml whole blood or 5 x 106 peripheral blood mononuclear cells.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1 - HIV Positive: Participant in parent study ATN 024, aged 12-24 years, testing HIV positive. All eligible youths must be negative for HBV core antibody, HBV surface antigen, and HBV surface antibody at the time of enrollment in to ATN 024.
- 2 - HIV Negative: Participant in parent study ATN 025, aged 12-24 years and testing negative for HIV infection. All eligible youths must be negative for HBV core antibody, HBV surface antigen, and HBV surface antibody at the time of enrollment in to ATN 025.

SUMMARY:
This laboratory-based substudy of an effectiveness trial of two Hepatitis B vaccines in HIV-negative youths is being done to evaluate the genetic contribution to the individualized immune response.

DETAILED DESCRIPTION:
This laboratory-based substudy of ATN 024 and 025 will evaluate the genetic contribution to highly individualized immune responses to hepatitis B vaccine in individuals and confirm the correlation of specific human leukocyte antigen (HLA) alleles and haplotypes with Hepatitis B Virus (HVB) antibody concentrations and antibody decay kinetics in vaccinated adolescents. Approximately 5 ml of whole blood will be collected from study participants at the time of the week 28 visit or at any subsequent study visit or clinic visit following successful completion of the week 28 visit. Peripheral blood mononuclear cells will be obtained and QIA amp Blood kit will be used to extract high-quality genomic DNA for polymerase chain reaction-based genotyping by the PEII laboratory.

The study is expected to be available for the duration of the parent studies which is approximately 2 years. This study requires one visit that may be arranged to coincide with a study or routine clinic visit. There are no follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Subjects currently enrolled in ATN 024 or ATN 025 are eligible for enrollment in ATN 052 beginning at or following completion of the week 28 visit.
* Subjects previously enrolled in ATN 024 or ATN 025 are eligible for enrollment in ATN 052, unless the subject was prematurely discontinued from the study prior to the first post-vaccination serology assessment which is performed at week 28.
* Current pregnancy is permitted.
* A signed informed assent/consent must be obtained from the subject.
* Written parental or guardian permission must be obtained where required by the institutional review board/ethics committee (IRB/EC).

Exclusion Criteria:

* Inadequate post-vaccination serology evaluation in ATN 024 or ATN 025.
* Unable to obtain informed consent and/or parental/legal guardian permission where required by the local IRB/EC.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All subjects who are currently enrolled or have completed ATN 024 or ATN 025 are eligible for participation on this substudy with the exception of those who were discontinued from ATN 024 or ATN 025 prior to completing the first post-vaccination serology (week 28) visit.
  Participants in ATN 024 are HIV-infected youths aged 12 to 24 years, while participants in ATN 025 are HIV-uninfected youths aged 12 to17 years, thus participants in this substudy will be HIV-infected and uninfected youth aged 12 to 24 years. All eligible youths must be negative for HBV core antibody, HBV surface antigen, and HBV surface antibody at the time of enrollment in to the parent protocols.
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To confirm the correlation of HLA-DRB1 and HLA-DQB1 alleles and haplotypes with HBV antibody concentrations and antibody decay kinetics in vaccinated adolescents. | Specimen obtained at or after the first post- vaccination serology visit.

SECONDARY OUTCOMES:
To determine if other genetic variations (768 single nucleotide polymorphisms (SNP) in about 50 genes) in the immune response pathways can confer additional effects on immune responses to hepatitis B vaccination. | Specimen obtained at or after the first post-vaccination serology visit.
To compare the strength of genetic and non-genetic associations with specific antibody responses following HBV vaccination. | Specimen obtained at or after the first post-vaccination serology visit.
To explore similarities and differences in genetic associations between HIV-positive and HIV-negative cohorts. | Specimen obtained at or after the first post-vaccination serology visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Tang, Ph.D, Study Chair — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Franciso, California
  - Children's Hospital National Medical Center, Washington D.C., District of Columbia
  - University of Southern Florida College of Medicine, Tampa, Florida

REFERENCES:
- See also: Adolescent Trials Network for HIV/AIDS Intervention — http://www.atnonline.org